CLINICAL TRIAL: NCT06419504
Title: The Effect of Ultrasonography-guided Pectoserratus Plane Block, Erector Spina Plane Block and Serratus Anterior Plane Block on Postoperative Opioid Consumption, Recovery Quality and Chronic Pain in Breast Cancer Surgery Patients
Brief Title: The Effect of Ultrasonography-guided Fascial Plane Blocks in Breast Cancer Surgery Patients
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 6/11
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: regional anesthesia; postoperative pain; recovery quality; chronic pain; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative; Chronic Pain | interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- SAP block group: Before the surgery, US-guided SAP block will be performed
  Interventions: Other: SAP block group
- PECS II block group: Before the surgery, US-guided PECS II block will be performed
  Interventions: Other: PECS II block group
- ESP block group: Before the surgery, US-guided ESP blockwill be performed
  Interventions: Other: ESP block group
- Control group: No intervention
  Interventions: Other: Control group

INTERVENTIONS:
Other: SAP block group — US-guided SAP block is performed approximately 30 minutes before the surgery in patients undergoing breast cancer surgery in a separate regional anesthesia room with standard anesthesia monitoring.
  Groups: SAP block group
Other: PECS II block group — US-guided PECS II block is performed approximately 30 minutes before the surgery in patients undergoing breast cancer surgery in a separate regional anesthesia room with standard anesthesia monitoring.
  Groups: PECS II block group
Other: ESP block group — US-guided ESP block is performed approximately 30 minutes before the surgery in patients undergoing breast cancer surgery in a separate regional anesthesia room with standard anesthesia monitoring.
  Groups: ESP block group
Other: Control group — No intervention
  Groups: Control group

SUMMARY:
The aim of this study was to evaluate the efficacy of serratus anterior plane (SAP) block, pectoserratus plane (PECS II) block, and erector spinae plane (ESP) block on postoperative acute pain, quality of recovery and chronic pain in breast cancer surgery patients.

DETAILED DESCRIPTION:
Breast cancer is the most common type of cancer in women. Although surgical treatment is effective and curative, it is associated with many complications in the postoperative period. Acute pain after surgery is one of them. Approximately half of women undergoing breast surgery describe significant post-operative pain (>5 on the Visual Analogue Scale; VAS) score that is not always effectively controlled by standard post-operative treatments. Poorly controlled postoperative pain has been associated with impaired functional recovery, delayed discharge from the post-anesthetic care unit, and prolonged hospital stay. In addition, poorly managed acute pain becomes chronic and is described as 'post-mastectomy pain syndrome'. Regional techniques can reduce acute and chronic postoperative pain. The development of ultrasonography (US)-guided regional anesthesia has led to the development of fascial plane blocks. Serratus anterior plan (SAP) block, pectoserratus plan (PECS II) block, and erector spina plan (ESP) block are frequently used for postoperative analgesia in patients undergoing breast surgery. he aim of this study was to evaluate the efficacy of serratus anterior plane (SAP) block, pectoserratus plane (PECS II) block, and erector spinae plane (ESP) block on postoperative acute pain, quality of recovery and chronic pain in breast cancer surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* elective breast surgery (modified radical mastectomy, breast conserving surgery, simple mastectomy, axillary lymph node dissection, etc.),
* 18 to 65 years old,
* American Society of Anaesthesiology (ASA) score I-III
* body mass index (BMI) <32 kg/m2

Exclusion Criteria:

* contraindications to the block applications
* history of mental or neurological disorders
* history of chronic opioid use
* chronic alcoholism
* substance use
* treatment of chronic pain
* severe liver and kidney disease
* uncooperative patients
* patients scheduled for bilateral mastectomy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The patients scheduled for elective breast surgery (modified radical mastectomy, breast conserving surgery, simple mastectomy, axillary lymph node dissection, etc.)
Study Population: It is planned to include ASA I-III patients between the ages of 18-65 who are planned to undergo breast cancer surgery
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2024-05-17 (Actual); Primary Completion 2024-09-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
postoperative opioid consumption | 24 hours
  All patients will receive a standard patient controlled analgesia (PCA) protocol. The postoperative opioid consumption will only be recorded.

SECONDARY OUTCOMES:
recovery quality | 5 minutes
  The Quality of Recovery-15 (QoR-15) is a 15-question questionnaire validated to assess poetoperative recovery. This questionnaire assesses patients' pain, physical comfort, physical independence, psychological support, and emotional status in the erly postoperative period. The patient is asked to express their status scoring from 0 to 10; therefore, the total score ranges from 0 to 150 points.
chronic pain | 3 months
  Patients will be telephoned 3 months after the operation and the presence, localization, and intensity of the pain, its character, and its relation with rest and/or activity will be recorded by asking only verbally.

CONTACTS AND LOCATIONS:
Overall Officials: Hafizenur O Atalay, M.D., Principal Investigator — University of Health Sciences, Antalya Training and Researh Hospital; Arzu O Karaveli, M.D., Principal Investigator — University of Health Sciences, Antalya Training and Researh Hospital
Locations (1):
- University of Health Sciences, Antalya Training and Researh Hospital, Antalya, Muratpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang S, Shi J, Dai Y, Zhang J, Liu Q, Yang P, Zhu N. The effect of different nerve block strategies on the quality of post-operative recovery in breast cancer patients: A randomized controlled study. Eur J Pain. 2024 Jan;28(1):166-173. doi: 10.1002/ejp.2178. Epub 2023 Sep 1. PMID 37655864
- [Background] Fujii T, Shibata Y, Akane A, Aoki W, Sekiguchi A, Takahashi K, Matsui S, Nishiwaki K. A randomised controlled trial of pectoral nerve-2 (PECS 2) block vs. serratus plane block for chronic pain after mastectomy. Anaesthesia. 2019 Dec;74(12):1558-1562. doi: 10.1111/anae.14856. Epub 2019 Sep 19. PMID 31535722